CLINICAL TRIAL: NCT05698238
Title: Phase Ib/ll Clinical Study to Evaluate Safety and Dosing of Humanised Monoclonal Antibody CA9hu-1 to Human Carbonic Anhydrase IX in Patients With Advanced Solid Tumours
Brief Title: Clinical Study to Evaluate Safety and Dosing of CA9hu-1 in Patients With Advanced Solid Tumours
Acronym: CAMP1
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mabpro, a.s. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MP01
Record Dates: First submitted 2023-01-04; First posted 2023-01-26 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Clear Cell Renal Cell Carcinoma Metastatic; TNBC - Triple-Negative Breast Cancer; Head and Neck Cancer; Non-small-cell Lung Carcinoma; Mesothelioma, Malignant
MeSH Terms: conditions — Clear-cell metastatic renal cell carcinoma; Triple Negative Breast Neoplasms; Head and Neck Neoplasms; Carcinoma, Non-Small-Cell Lung; Mesothelioma, Malignant

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment arm (Experimental)
  Interventions: Drug: CA9hu-1

INTERVENTIONS:
Drug: CA9hu-1 — Humanized monoclonal antibody to human carbonic anhydrase IX

SUMMARY:
Carbonic anhydrase IX (CA IX) has been implicated in the progression of most solid tumours and expression has been demonstrated in clinical samples from a variety of solid cancers. High expression is often associated with high grade or metastatic disease and poor prognosis. CA IX is not expressed in normal tissue, potentially providing a cancer-associated target that would not likely result in significant interruption of normal biologic function in organs not affected by cancer. A humanized monoclonal antibody CA9hu-1 has shown robust activity in a variety of tumour models including models of ovarian, prostate, breast, pancreatic, colon and lung where tumour growth and metastasis are inhibited when CA9hu-1 is used as a monotherapy. Enhancement of chemotherapy has also been demonstrated in several models in combination with CA9hu-1. CA IX is also expressed by tumour-associated cells (angiogenic endothelium, tumour-associated macrophages), which also drive cancer progression. Thus, targeting CA IX with CA9hu-1 in cancer patients is expected to affect multiple pathways and multiple tumour compartments that are important to tumour progression. Taken together, there is strong rationale for developing hu-CA91 for the treatment of advanced cancer. The present study was designed to establish safety and toxicity profile and maximum tolerated dose of CA9hu-1, evaluate pharmacokinetics, investigate the presence of anti-drug antibody, to document anti-tumour activity at a clinically relevant dose, and to document the use of [18F]FLT-PET as a biomarker for detection of early tumour response at a clinically relevant dose.

ELIGIBILITY:
Inclusion Criteria:

* Written (signed and dated) informed consent and be capable of co-operating with treatment and follow-up
* Histologically proven solid tumors (Clear Cell Renal Cell Carcinoma Metastatic, Triple-Negative Breast Cancer, Head and Neck Cancer, Non-small-cell Lung Carcinoma, Malignant Mesothelioma) refractory to conventional treatment, or for which no conventional therapy is considered appropriate by the Investigator or is declined by the patient
* Life expectancy of at least 12 weeks
* World Health Organization (WHO) performance status of 0 or 1
* Hematological and biochemical indices within the ranges (hemoglobin ≥9.0 g/dL, absolute neutrophil count ≥1.5 x 109/L, platelet count ≥100 x 109/L, bilirubin ≤1.5 x upper limit of normal, alanine amino-transferase (ALT) and aspartate amino-transferase (AST) ≤ 2.5 x upper limit of normal. These measurements must be performed within one week (Day -7 to Day -1) before the patient receives their first infusion of CA9hi-1.
* Calculated creatinine clearance or isotope clearance measurement ≥ 50 mL/min
* PT/APTT ≤1.5 upper limit of normal

Exclusion Criteria:

* Ongoing toxic manifestations of previous treatments (Grade 2 or greater according to NCI-CTCAE v4.02) with the exception of alopecia or certain Grade 2 toxicities, which in the opinion of the investigator and CDD should not exclude the patient - these should be discussed on a case by case basis
* Symptomatic brain metastases or spinal cord compression
* Patients who have received prior radiotherapy to their lungs will not be eligible for this trial.
* Female patients who are able to become pregnant (or already pregnant or lactating). However, those patients who have a negative serum or urine pregnancy test before enrolment and agree to use two highly effective forms of contraception (oral; injected or implanted hormonal contraception and condom; have an intra-uterine device and condom; diaphragm with spermicidal gel and condom) effective at the first administration of CA9hu-1, throughout the trial and for six months afterwards are considered eligible. Breast feeding should be discontinued if the mother is treated with CA9hu-1.
* Male patients with partners of child-bearing potential (unless they agree to take measures not to father children by using one form of highly effective contraception [condom plus spermicide] effective at the first administration of hu-CA91, throughout the trial and for six months afterwards). Men with pregnant or lactating partners must be advised to use barrier method contraception (for example: condom plus spermicidal gel) to prevent exposure to the foetus or neonate.
* Any major surgical procedure within 4 weeks prior to patients scheduled Cycle 1 Day 1, any major thoracic or abdominal surgery from which the patient has not yet recovered.
* A serious or non-healing active wound, ulcer, or bone fracture.
* At high medical risk because of non-malignant systemic disease including active uncontrolled infection.
* Known to be serologically positive for Hepatitis B, Hepatitis C or Human Immunodeficiency Virus (HIV) or who have an active, ongoing infection or an active, known or suspected autoimmune disease or on systemic steroids.
* Concurrent congestive heart failure, prior history of class III/ IV cardiac disease (New York Heart Association [NYHA]), prior history of cardiac ischemia or prior history of cardiac arrhythmia.
* Is a participant or plans to participate in another interventional clinical trial, whilst taking part in this Phase I study of CA9hu-1. Participation in an observational trial or interventional clinical trial which does not involve administration of an IMP and which would not place an unacceptable burden on the patient in the opinion of the Investigator and Medical Advisor would be acceptable.
* Any other condition which in the Investigator's opinion would not make the patient a good candidate for the clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events to CA9hi-1 and grading their severity according to the National Cancer Institute's Common Terminology Criteria for adverse Events (NCI CTCAE) Version 4.02. | 6 months
  The primary objective of this outcome is to establish the safety and toxicity profile of hu-CA91.
Number of patients reaching the dose levels of 750 mg of CA9hu-1 without any dose limiting toxicities. | 4 weeks
  The objective of this outcome is to perform a dose escalation of of CA9hu-1 to levels of 750mg without any dose limiting toxicities.
Number of patients reaching pharmacologically active dose measurement of CA9hu-1 | 4 weeks
  The objective of this outcome is to determine number of patients in whom the pharmacologically active dose of CA9hu-1 wil be reached by measurement of plasma concentrations of the CA9hu-1. In order to reach the proposed pharmacologically active dose, the plasma levels of 200 +/- 100 nM are necessary.
Maximum tolerated dose of CA91hu-1 | 4 weeks
  The objective is to determine a dose at which no more than one patient out of up to six patients at the same dose level experience a highly probable or probable CA9hu-1 related dose limiting toxicity.

SECONDARY OUTCOMES:
Half-life of CA9-hu-1 | 4 weeks
  Measurement of CA9hu-1 half-life after human administration provides basic PK descriptive data.
Peak Plasma Concentration (Cmax) of CA9hu-1 | 4 weeks
  The measurement of Cmax after CA9hu-1 administration will provide basic PK descriptive parameter of the drug.
Area under the plasma concentration versus time curve (AUC) | 4 weeks
  The measurement of AUC after CA9hu-1 administration will provide basic PK parameter of the drug.
Anti-drug antibodies | 6 months
  Analyses of plasma samples for presence of anti-drug antibodies following CA9hu-1 administration
Anti-tumour activity of CA9hu-1 | 6 months
  Evaluate response (stable disease, partial response or complete response) in any of the patients as determined by the Response Evaluation Criteria in Solid Tumours Version 1.1 (RECIST).
Biomarker for detection of early tumour response | 6 months
  Determination of the magnitude of change in apparent standard uptake volume (SUV) calculated from the uptake of FLT by tumour tissue quantified by [18F]FLT-PET during the second cycle of CA9hu-1 treatment and the relation with response

IPD SHARING:
Plan to Share IPD: Undecided